CLINICAL TRIAL: NCT05532423
Title: Effect of Nitrate Supplementation on Cerebrovascular Function and Cognitive Function in Older Adults With Metabolic Syndrome
Brief Title: Nitrate Supplementation and Cerebrovascular and Cognitive Function in Metabolic Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David N. Proctor, PhD, Principal Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00020830
Record Dates: First submitted 2022-08-26; First posted 2022-09-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Syndrome
Keywords: Cognition
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The design is a single group randomized crossover trial, with individuals with metabolic syndrome receiving both the active nitrate rich juice and the placebo juice, randomized in order.
Who Masked: Participant, Investigator
Masking Description: As it is a double blind study, participants and investigators for this study will be blinded to the intervention they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metabolic Syndrome Older Adult (Experimental): Participants with metabolic syndrome will be drinking nitrate rich beetroot juice from the James White Beet It company. Participants will drink one dose of 140mL beetroot juice for two visits of either a nitrate rich juice or a nitrate depleted placebo drink. Both drinks taste and smell the same, just with the active component removed. Following these visits, participants will drink 70ml of nitrate rich beetroot juice daily for 4 weeks to investigate long term effects of the juice on study outcomes.
  Interventions: Drug: Beetroot Juice - Active
- Metabolic Syndrome Older Adult - Placebo juice condition (Experimental): Participants with metabolic syndrome will be drinking nitrate rich beetroot juice from the James White Beet It company. Participants will drink one dose of 140mL beetroot juice for two visits of either a nitrate rich juice or a nitrate depleted placebo drink. Both drinks taste and smell the same, just with the active component removed. Following these visits, participants will drink 70ml of nitrate rich beetroot juice daily for 4 weeks to investigate long term effects of the juice on study outcomes.
  Interventions: Drug: beetroot juice - Placebo

INTERVENTIONS:
Drug: Beetroot Juice - Active — Participants with Metabolic syndrome will drink 140mL of organic nitrate rich beetroot juice from the James White Beet It Company. This juice will be the active juice, meaning it has the high nitrate content that is of interest. This drink will be given two 70 mL bottles of the juice that will be blinded to them and investigators.
  Other Names: Experimental
  Arms: Metabolic Syndrome Older Adult
Drug: beetroot juice - Placebo — Participants with Metabolic syndrome will drink 140mL of organic nitrate rich beetroot juice from the James White Beet It Company. This drink will be the placebo drink, which means all of the nitrate has been extracted, however it tastes and smells the same as the active drink. This drink will be given two 70 mL bottles of the juice that will be blinded to them and investigators.
  Other Names: Placebo
  Arms: Metabolic Syndrome Older Adult - Placebo juice condition

SUMMARY:
The purpose of this study is to determine if beetroot juice consumption can improve cognitive performance and brain vascular function in individuals with metabolic syndrome

DETAILED DESCRIPTION:
Metabolic syndrome is a preclinical state that is related to increased risk of cardiovascular and metabolic disease. The purpose of this study is to determine if beetroot juice consumption can improve cognitive performance and brain vascular function in individuals with metabolic syndrome. The first part of this study will aim to determine if people with metabolic syndrome present with poorer brain vascular function and cognitive performance relative to older adults without metabolic syndrome. The second part of this study aims to determine whether brain vascular functions and cognitive function can be improved with beetroot juice.

Cognitive function is highly related to the ability of the brain to deliver blood to specific regions of the brain. The brain has many blood vessels and relies on a healthy and intact vascular system to optimally perform. With aging and disease risk factors that relate to metabolic syndrome, cognition and brain function and structure decline at a more rapid pace. These changes may directly impact quality of life, financial burden, and independence. Therefore, determining the cognitive and brain functional changes that occur due to metabolic syndrome is an important clinical and scientific question.

This research study will assess whether dietary nitrate, in the form of beetroot juice, can improve brain blood vessel function and cognition in adults with metabolic syndrome. Beetroot juice has a high content of dietary nitrate, which has known beneficial effects on blood vessel function and blood pressure. With aging and disease risk factors, you lose the ability to dilate the blood vessels, reducing how much blood can get to the brain. Providing dietary nitrate in the form of beetroot juice may help improve blood vessel dilation and cognitive function in individuals with metabolic disease risk factors. Additionally, intervening during metabolic syndrome, before disease progresses to cardiovascular disease and diabetes, is optimal to minimize the long-term effects on cognition and brain health.

ELIGIBILITY:
Inclusion Criteria:

MetS classification according to NCEP III definition - MetS group only … at least 3 of the 5 components Individuals with a waist circumference >102 cm (40 in) for men > 88 cm for women Triglycerides ≥150 mg/dL HDL cholesterol ≤ 50 mg/dL for women and ≤ 40 mg/dL for men Blood pressure ≥130/85 mmHg Fasting blood glucose ≥100 mg/dL Age 55-75 Men and women All races and ethnicities

Exclusion Criteria:

1. Individuals with any overt cardiovascular, hematologic, pulmonary, renal, musculoskeletal, and/or neurological disease(s).
2. Premenopausal women - indicated by mention of last menstrual cycle
3. Individuals with active cancer
4. Individuals with moderate/severe depressive disorder as indicated by BDI-II scores (BDI-II score >14)
5. Individuals with cognitive impairment as indicated by the MMSE (score on the MMSE < 24)
6. Individuals with visual impairment
7. Users of any tobacco and/or nicotine products (smokers, chewing tobacco, nicotine-containing patches/gum, smokeless cigarettes)
8. Individuals taking hormone replacement
9. Taking following an of the following medications:

   1. nitrates (e.g. nitroglycerin) for angina
   2. phosphodiesterase inhibitors (e.g., Viagra)
   3. anti-Inflammatory drugs

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Functioning - Change in N-back test performance | At Baseline, 90 minutes following drinking the beetroot juice (single 140mL acute dose), 90 minutes following drinking the placebo drink (single 140mL acute dose), and after 4 weeks of daily (70mL) beetroot juice consumption
  Reaction time of responses for each trial type (0-back, 1-back, 2-back, and 3-back)
Cognitive Functioning - Change in N-back test performance | At Baseline, 90 minutes following drinking the beetroot juice (single 140mL acute dose), 90 minutes following drinking the placebo drink (single 140mL acute dose), and after 4 weeks of daily (70mL) beetroot juice consumption
  Percent accuracy of correct responses for each trial type (0-back, 1-back, 2-back, and 3-back)
Changes in Cerebral Autoregulation - NIRx (fNIRS/cerebral oxygenation) and finapres (blood pressure) derived waveforms for transfer function analysis | At Baseline, 90 minutes following drinking the beetroot juice (single 140mL acute dose), 90 minutes following drinking the placebo drink (single 140mL acute dose), and after 4 weeks of daily (70mL) beetroot juice consumption
  This outcome will be measured using non-invasive methodology utilizing fNIRS and will involve rhythmic breathing to determine the relation between blood pressure and an index of blood flow. The variable of interest is the phase derived from transfer function analysis of the blood pressure and fNIRS waveforms.
Changes in Neurovascular Coupling - changes in fNIRS signals during the N-back cognitive test | At Baseline, 90 minutes following drinking the beetroot juice (single 140mL acute dose), 90 minutes following drinking the placebo drink (single 140mL acute dose), and after 4 weeks of daily (70mL) beetroot juice consumption
  This outcome will also be measured using fNIRS and will involve measurement of brain oxygenation during cognitive assessment. The variable of interest will be changes in fNIRS oxyhemoglobin and deoxyhemoglobin signals (% change from baseline) during the cognitive assessment (n-back test).

SECONDARY OUTCOMES:
Changes in Pulse Wave Velocity - Colin Cardiovascular Profiling System 2000 | At Baseline, 90 minutes following drinking the beetroot juice (single 140mL acute dose), 90 minutes following drinking the placebo drink (single 140mL acute dose), and after 4 weeks of daily (70mL) beetroot juice consumption
  Participants will have arterial stiffness (cm/s) assessed at certain time points to determine if beetroot juice impacts this outcome
Taste Profile of Juice (Sweetness, Bitterness, and Sourness) - Questionnaire developed in our lab | This will be taken one time, at the last study visit after 4 weeks of juice consumption
  A survey questionnaire will be used to characterize participants perception and thoughts on the beetroot juice which will help determine the potential clinical translation of beetroot juice in this population. This scale will be 1-10 and a higher score indicates more of that taste.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, Noll Lab, University Park, Pennsylvania, United States